CLINICAL TRIAL: NCT01576302
Title: Diaphragmatic Breathing and Progressive Muscle Relaxation: Behavioral Interventions for Gastrointestinal Rumination
Brief Title: Comparison of Diaphragmatic Breathing and Muscle Relaxation for Rumination
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Richard J. Seime, PHD, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11-008528
Record Dates: First submitted 2012-04-09; First posted 2012-04-12 (Estimated); Last update posted 2014-12-10 (Estimated); Status verified 2014-12

CONDITIONS: Rumination
Keywords: Rumination
MeSH Terms: conditions — Rumination Syndrome | interventions — Muscle Relaxation; Relaxation Therapy; Autogenic Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Diaphragmatic breathing (Experimental): Training in diaphragmatic breathing as response incompatible with rumination.
  Interventions: Behavioral: Diaphragmatic breathing; Behavioral: Muscle relaxation
- Muscle relaxation (Active Comparator): Patients in this arm of study will be taught muscle relaxation as intervention for rumination, instructed in habit-reversal paradigm to use after eating food or if urge to ruminate
  Interventions: Behavioral: Muscle relaxation

INTERVENTIONS:
Behavioral: Diaphragmatic breathing — Patients in this arm will be provided training in diaphragmatic breathing, taught its application in habit-reversal paradigm (to use after eating food and if urge to ruminate).
  Arms: Diaphragmatic breathing
Behavioral: Muscle relaxation — Progressive passive muscle relaxation
  Other Names: Relaxation training; Progressive Muscle Relaxation

SUMMARY:
Rumination is an upper gastrointestinal (GI) disorder characterized by the frequent regurgitation of recently ingested food. Very little is understood about the nature and treatment of this disorder. The act of regurgitation in rumination involves the opening of the upper esophageal sphincter and the muscular contraction of the abdomins rectus. Behavioral treatment of these symptoms is the clinical intervention of choice; however, only uncontrolled case documentation exists to support its effectiveness. However, an effective behavioral mechanism may be relaxation of the muscles. From a behavioral standpoint, muscular relaxation is incompatible with the necessary muscular contraction for rumination.

To date, single case documentation and few designed single case studies have examined the clinical effectiveness of behavioral interventions for GI rumination. In the current study, the investigators seek to examine the effectiveness of two behavioral relaxation interventions for GI rumination through a treatment as usual paradigm (proposed N = 20). Our primary goals are to examine the clinical effectiveness of these interventions in symptom reduction at 1- and 3-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years of age.
2. Diagnosis of rumination by RomeIII criteria

Exclusion Criteria:

1. Active alcohol or substance abuse
2. Presence of a depressive disorder as measured by PHQ-9 score of 10 or above
3. Presence of clinical significant anxiety disorder as measured by GAD-7 score of 10 or above.
4. Severe levels of health focused anxiety as measured by SHAI score of 26 or above.
5. Any medical, neurological, or psychiatric condition that would impair the ability to consent and carry out all study procedures.
6. Any active psychosis or suicidality.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2012-04; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Rumination Frequency assessed using Rome III Criteria | 1 month after intervention
  Study participants will be treated with diaphragmatic breathing in one arm and muscle relaxation in the other arm. Outcome measure is:
  Rome III Study Questions
  Q8: In the last week, how often did food come back up into your mouth?
  Q10: When food came back up into your mouth, did it usually stay in your mouth for a while before you swallowed it or spit it out?
Rumination frequency assessed using Rome III Criteria | 3 months after intervention
  Study participants will be treated with diaphragmatic breathing in one arm and muscle relaxation in the other arm. Outcome measure is:
  Rome III Study Questions
  Q8: In the last week, how often did food come back up into your mouth?
  Q10: When food came back up into your mouth, did it usually stay in your mouth for a while before you swallowed it or spit it out?

SECONDARY OUTCOMES:
Heath Care Utilization | 1 month after intervention
  How many healthcare visits would you estimate were related to rumination since you started the intervention?
Short Health Anxiety Inventory (SHAI) | 1 month post intervention
  Measure of degree to which intervention has impacted health concerns/anxiety. The SHAI is a validated measure
Sheehan Disability Scale (SDS) | 1 month after intervention
  This is a measure of the impact of symptoms on Work, Family, and Social life. Uses a 10 point scale --with categories of mild,moderate severe
Treatment adherence | 1 month after intervention
  Following question will be posed: Did you engage in the intervention as you were instructed at your training session? The responses will be categorized for themes.
Heath Care Utilization | 3 month after intervention
  How many healthcare visits would you estimate were related to rumination since you started the intervention?
Short Health Anxiety Inventory (SHAI) | 3 months post intervention
  Measure of degree to which intervention has impacted health concerns/anxiety. The SHAI is a validated measure
Sheehan Disability Scale (SDS) | 3 months after intervention
  This is a measure of the impact of symptoms on Work, Family, and Social life. Uses a 10 point scale --with categories of mild,moderate severe
Treatment adherence | 3 months after intervention
  Following question will be posed: Did you engage in the intervention as you were instructed at your training session? The responses will be categorized for themes.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Seime, PhD, LP, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States